CLINICAL TRIAL: NCT06795919
Title: Use of Particulate Cortico- Cancellous Anterior Iliac Graft with Periosteal Membrane in Treatment of Unilateral Alveolar Cleft Grafting Versus Particulate Cortico-cancellous Anterior Iliac Grafting Alone a Randomized Clinical Trial
Brief Title: Use of Particulate Cortico- Cancellous Anterior Iliac Graft with Periosteum Membrane in Unilateral Alveolar Cleft Grafting Versus Particulate Cortico-cancellous Anterior Iliac Grafting Alone.
Acronym: periosteum
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nesma Mattar (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Nesma Mattar, PHD candidate at Cairo University. Lecturer Assistant of Oral and Maxillofacial Surgery in New Giza University., Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bone graft in alveolar cleft
Record Dates: First submitted 2025-01-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Bone Grafting
Keywords: alveolar cleft; alveolar cleft bone graft; periosteum membrane; anterior ilium bone graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- secondary surgical repair of alveolar cleft with cortico-cancellous anterior iliac bone graft. (Experimental): The cleft area is infiltrated with 1% xylocaine with epinephrine on the palatal and buccal side of the anterior maxilla. Two full thickness mucoperiosteal flaps are created by incising the anterior surface of the alveolar process, alongside the cleft ridge. The nasal mucosa is separated by an incision from the gingiva on both sides of maxilla. Flaps are lifted cautiously with a periosteal elevator along the labial surface of alveolar process to the piriform aperture. The nasal mucosa is reflected into the nose and the periosteum out of the cleft so that new bone can be grafted. The autogenic bone fills the cleft fissure, and it is covered with lifted flaps. The incision of mucous flap for covering clefts can be moved from the lateral sides of the alveolar process. It is advised to place the bone graft in the region of the piriform aperture to provide elevation and support for the base of ala nasi on the cleft. The skin incision line is made parallel to the iliac crest.
  Interventions: Procedure: : delayed surgical repair of alveolar cleft using particulate cortico-cancellous anterior iliac bon

INTERVENTIONS:
Procedure: : delayed surgical repair of alveolar cleft using particulate cortico-cancellous anterior iliac bon — skin incision was marked 2-4 cm from the crest to anterior iliac spine height. This is done to avoid pain at the beltline if the incision is made directly over the anterior ilium. As well as avoid injury to the lateral femoral cutaneous nerve. After the anatomical marking are drawn using betadine solution, the site is injected with local anesthesia at the subcutaneous level. The skin incision line is made parallel to the iliac crest and posterior to the anterior iliac spine. Scalpel blade number 10 is used. The incision of the skin and subcutaneous fat was performed. Blunt dissection is carried out at the level of subcutaneous tissues to separate the fascia from fat. Cautery is used to control any hemorrhage. Using a number 15 blade, fascia was incised which covers the iliac spine. A hypo vascular plane was identified. It is located over the anterior iliac spine, as well as between the insertions of tensor fascia laterally and the external and the transverse abdominal muscles medially

SUMMARY:
In the past few years, periosteal membrane has been used in orthopedic surgery as well as periodontal surgery as a mechanism to promote bone healing without the ingrowth of fibrous tissues. It has shown its efficiency in maintaining the bone volume and density in postoperative follow up. This can in turn solve the problem of potential bone loss in patients of alveolar cleft.

The study aims to see if fixing the periosteum of the anterior ilium with tacks after bone graft application in the donor site will help maintain the graft and promote healing for the alveolar cleft patients

DETAILED DESCRIPTION:
Cleft lip and palate are the most common congenital deformity affecting craniofacial structures. Delayed alveolar cleft defect presents a challenge for reconstruction to achieve functional and esthetic results. Many sources of bone graft have been shown in the literature: cortical or cancellous bone, iliac crest, cranial bone, mandibular symphysis, tibia, and rib. The main complication is graft loss partial or complete and/or fistula formation postoperative.

Periosteal membrane was reported to be used in a comparative study in rabbits versus that of resorbable collagen membrane to assess iliac bone graft resorption. The results seem promising. Periosteum as a membrane shows superior reparative powers.

In the past few years, periosteal membrane has been used in orthopedic surgery as well as periodontal surgery as a mechanism to promote bone healing without the ingrowth of fibrous tissues. It has shown its efficiency in maintaining the bone volume and density in postoperative follow up. This can in turn solve the problem of potential bone loss in patients of alveolar cleft.

The study aims to see if fixing the periosteum of the anterior ilium with tacks after bone graft application in the donor site will help maintain the graft and promote healing for the alveolar cleft patients.

The most common cause of poor lifestyle, speech and feeding for secondary alveolar cleft patient is the communication of the oral cavity with the nasal cavity. Radiation, teratogenic drugs, nutritional deficiency, chemical exposure, and maternal hypoxia are all predisposing factor to the incidence an infant developing cleft.

The main aims in reconstruction surgery are to achieve complete anatomical and functional seal to obtain normal speech, without regurgitation of fluids or food into the nasal cavity. Another goal is to allow for normal maxillary growth. Fistula occurring has high incidence in appearing postoperative to the reconstruction surgery. This leads to future difficult management. Another possible complication is wound dehiscence and graft exposure.

Several studies attempted to resolve the complications with different bone graft sources whether autogenous, xenograft or allograft. The literature shows the use of different membranes to preserve the graft such as: PRF, collagen membrane and pericardium or completely without.

The main objective for conducting this research is to check if the usage of periosteum of the same donor site of the anterior ilium will in fact preserve the bone graft volume and density of the known gold standard graft and prevent possible complications.

The Periosteal flap stretch with fixation using tacks overlying the bone graft in cleft patients. It will be compared to using the gold standard corticocancellous graft without use of periosteal membrane.

Periosteum is a specialized connective tissue forming a thin and fibrous membrane firmly anchored to bone. In children, it is thicker, more vascular, and more loosely attached. It has high bone forming potential. Many studies show that periosteum regenerates both bone and cartilage.

The periosteum consists of two layers; the outer layer containing fibroblasts, vessels and sharpey's fibers. The inner layer contains undifferentiated mesenchymal cells, capillaries, and osteoblasts. This induces hematoma followed by callus formation during healing as it triggers sequences of cellular and biochemical events.

ELIGIBILITY:
Inclusion Criteria:

* 9 -12 years, depending on dental age not chronological.
* systemically healthy patients (American Society of Anesthesiologists -ASA I and II)
* Patients secondary alveolar cleft patient.

Exclusion Criteria:

* Patients with recurrent palatal fistula.
* Existence of syndromic cleft palate.
* Patient with uncontrolled systematic disease.
* Patients undergoing radiotherapy or chemotherapy for malignancy.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bone gain | 0-6 months
  CBCT , measured in cm
Bone Density | Preoperative, 1week postoperative & sixth months.
  CBCT , measured in Hounsfield units.

SECONDARY OUTCOMES:
Pain at Donor site | Immediate postoperative. 6 months
  Visual Analogue scale from 0 to 10.
Pain at Recipient site | Immediate postoperative. 6 months
  Visual Analogue scale from 0 to 10.
Infection | Immediate postoperative
  Yes/no
Patient satisfaction | Immediate postoperative and 6months.
  Yes/NO
Wound healing at donor and recipient site | Immediate postoperative. 6 months
  Clinical photos

CONTACTS AND LOCATIONS:
Overall Officials: Tarek El faramawi, Lecturer of OMFS, Study Chair — Cairo University
Locations (1):
- School of Dentistry, Cairo., Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Shahba AG, Wilkman T, Kornilov R, Adam M, Salla KM, Linden J, Lappalainen AK, Bjorkstrand R, Seppanen-Kaijansinkko R, Mannerstrom B. Periosteal Flaps Enhance Prefabricated Engineered Bone Reparative Potential. J Dent Res. 2022 Feb;101(2):166-176. doi: 10.1177/00220345211037247. Epub 2021 Sep 11. PMID 34514892